CLINICAL TRIAL: NCT00644345
Title: Reproducibility of T Wave Alternans Testing in Patients With Ischemic Heart Disease.
Brief Title: T-Wave Alternans (TWA) Reproducibility in CAD Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Therese Fuchs, MD, Assaf Harofeh Medical Center
Other Study IDs: 38-08
Record Dates: First submitted 2008-03-23; First posted 2008-03-26 (Estimated); Last update posted 2008-03-26 (Estimated); Status verified 2008-03

CONDITIONS: Coronary Artery Disease
Keywords: Microvolt T wave alternans; reproducibility
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Microvolt T-Wave Alternans (MTWA) is a relatively new non-invasive method for identifying patients at increased risk of sudden death from ventricular arrhythmias. MTWA can be measured during a routine exercise test, during pharmacologic stress or during cardiac pacing. Its clinical performance compares favorably with that of other non-invasive risk stratifiers and invasive electophysiologic studies. The purpose of the present study is to define the reproducibility of MTWA testing.

DETAILED DESCRIPTION:
The study will be performed in the Cardiac Rehabilitation Center at Assaf Harofeh Medical Center. Patients with coronary artery disease will be eligible to enroll.

Patient will undergo an exercise test on a stationary bicycle. TWA will be measured at heart rate of 105 and 115 BPM. The test will be repeated one week later in the same fashion. The patient will continue follow-up in the rehabilitation center as dictated by the rehabilitation program. Patients will be kept on their regular medications and there will be no change of the medications from the first TWA measurement to the second.

ELIGIBILITY:
Inclusion Criteria:

1. Patients enrolled in the cardiac rehabilitation center program
2. Patients with CAD
3. Age >18 and < 80 YO
4. Patients with a pacemaker or defibrillator with normal AV conduction

Exclusion Criteria:

1. Patients with chronic AF
2. Patients with multiple APB's or PVC's
3. Patients who are unable to increase their heart rate to 115 BPM and don't have a pacemaker.
4. Patients who are unable to exercise on a bicycle.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease enrolled in a cardiac rehabilitation program.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-01 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Reproducibility of TWA test results | 1 week

SECONDARY OUTCOMES:
Ventricular arrhythmias during exercise | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Therese Fuchs, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Assaf Harofeh Medical Center, Zrifin, Israel